CLINICAL TRIAL: NCT00277927
Title: Clinical Management of Children With Mild Valvar Pulmonary Stenosis
Brief Title: Mild Valvar Pulmonary Stenosis
Status: Terminated | Type: Observational
Why Stopped: sufficient data collected for significant study results
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: William T Mahle, MD, Children's healthcare of Atlanta
Other Study IDs: 04-035
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2007-11

CONDITIONS: Congenital Disorders
Keywords: Pediatric; Cardiac; Valvar Pulmonary Stenosis
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Pulmonary Valve Stenosis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Mild valvar pulmonary stenosis can be detected in 1/10,000 live births. Historical data suggested that most of these patients do well. Nonetheless, the majority of these patients is followed periodically by a pediatric cardiologist and may undergo repeated echocardiographic studies to follow the gradient. Such follow-up can be costly and it is not know if there is any benefit to periodic evaluation.

DETAILED DESCRIPTION:
Young children (less than or equal to 2 years of age) with mild valvar pulmonary stenosis are unlikely to develop worsening stenosis with age and periodic cardiac evaluation is not warranted.

To describe the clinical course of children with mild valvar pulmonary stenosis diagnosed in early childhood. To examine the clinical practice patterns of cardiologists caring for these patients.

Retrospective chart review of all children diagnosed with mild valvar pulmonary stenosis born between 1984 and 2003 and followed by Sibley Heart Center Cardiology. Patient variables will include: pulmonary valve gradient, need for catheterization, exercise intolerance and endocarditis. Practice variables will include: frequency of follow-up, number of echocardiographic studies, exercise limitations.

ELIGIBILITY:
Inclusion Criteria:

* Children's Healthcare of Atlanta medical charts 1984 to 2003 diagnosed with mild valvar pulmonary stenosis Patients less than or equal to two years of age

Exclusion Criteria:

* Those who do no meet inclusion criteria

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children at Children's Healthecare of Atlanta between the dates of 1984 and 2003 with mild valvar pulmonary stenosis that were less than 2 years old
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 1984-01; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T. Mahle, MD, Principal Investigator — Children's Healthcare of Atlanta, Sibley Heart Center Cardiology
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States